CLINICAL TRIAL: NCT01985451
Title: Phase II Trial of Pemetrexed and Temozolomide in Treating Patients With Relapsed PCNSL
Brief Title: Pemetrexed and Temozolomide in Treating Patients With Relapsed Primary Central Nervous System Lymphoma （PCNSL）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rongjie Tao (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Rongjie Tao, Neurosurgery, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI002; ShandongCHI (Registry Identifier: ShandongCHI)
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Central Nervous System Tumors
Keywords: Lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma | interventions — Pemetrexed; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed and Temozolomide (Experimental): Patients with relapsed PCNSL patients were treated with high-dose pemetrexed (900mg/m2) and temozolomide (200mg/m² day 1-5, 28 day cycle).
  Interventions: Drug: Pemetrexe; Drug: Temozolomide

INTERVENTIONS:
Drug: Pemetrexe — Patients with relapsed PCNSL patients were treated with high-dose pemetrexed (900mg/m²).
  Other Names: Alimta
Drug: Temozolomide — Patients with relapsed PCNSL patients were treated with temozolomide (200mg/m² day 1-5,28).
  Other Names: Temodal

SUMMARY:
In this trial, we will treat relapsed PCNSL with temozolomide, pemetrexed. Our objective was to assess our treatment strategies' availability based on response rates, progression-free survival (PFS), median PFS, and toxicity.

DETAILED DESCRIPTION:
The best reported outcomes of PCNSL treatment are high-dose methotrexate-based chemotherapy combined with whole-brain radiation therapy (WBRT). Despite aggressive therapy, however, nearly 50% of patients will relapse within 24 months of diagnosis. Furthermore, the application of high-dose methotrexate-based regimen is complex, needing be hydrated, alkalified and detoxified, and treatment-related toxicity mortality is severe. In an attempt to improve upon these poor results and reduce treatment-related side effects, we will treat about 15-20 relapsed PCNSL patients who was fail in high-dose methotrexate-based chemotherapy. Our objective is to assess our treatment strategies' availability based on response rates, progression-free survival (PFS), median PFS, and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary CNS lymphoma.
* ECOG (Eastern Cooperative Oncology Group) Performance status of 0-1.
* Positive cerebrospinal fluid (CSF) cytology or immunohistochemical diagnosis of CSF monoclonality with or without measurable intracranial disease.
* Measurable (greater than 1 cm in diameter) tumor by CT scan or MRI.
* Progressed during first-line chemotherapy and/or radiotherapy OR relapsed after initial successful treatment.
* No systemic lymphoma by CT scan of the chest, abdomen, and pelvis with contrast.
* No leptomeningeal lymphoma by lumbar puncture for CNS cytology/flow cytometry.
* No ocular lymphoma by slit lamp examination.
* Must have adequate organ function as defined by the protocol: Adequate renal function: serum creatinine ≤ 1.5 mg/dl and/or calculated creatinine clearance ≥ 60 ml/min; Adequate hepatic function: bilirubin level ≤ 1.5 x ULN, ASAT & ALST ≤ 1.5 x ULN.Adequate bone marrow reserves: neutrophil (ANC) count ≥ 1500 /mm^3, platelet count ≥ 100,000 /mm^3, hemoglobin ≥ 9 g/dl.
* Age >/= 18 and </= 75 years.
* Signed written informed consent prior to study entry.

Exclusion Criteria:

* Patients with human immunodeficiency virus seropositivity and systemic lymphoma manifestation.
* Serious uncontrolled concurrent illness.
* Previous brain radiotherapy, systemic chemotherapy.
* Concurrent chronic systemic immune therapy, targeted therapy not indicated in this study protocol.
* Any evidence of prior exposure to Hepatitis B virus.
* Unable to comprehend the study requirements or who are not likely to comply with the study parameters.
* Pregnant (confirmed by serum or urine β-HCG) or lactating.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) | 2 years
  Contrast MRI was performed to assess treatment response at 3-month interval for 2 years and thereafter every 6 months for next 3-5 years and then annually. The treatment response was reassessed according to International PCNSL Collaborative Group' criteria[1].
  [1] Abrey LE, Batchelor TT, Ferreri AJ, Gospodarowicz M, Pulczynski EJ, Zucca E, et al. Report of an international workshop to standardize baseline evaluation and response criteria for primary CNS lymphoma. International Primary CNS Lymphoma Collaborative Group. J Clin Oncol 2005;23:5034-43.

SECONDARY OUTCOMES:
Failure-free survival (PFS) | 2 years
  Contrast MRI was performed to assess treatment response. PFS was defined as the time from initial diagnosis until disease progression. PFS and median PFS were analyzed using the Kaplan-Meier product limit curve.
Toxicity | 2 years
  Toxicity was graded according to the Word Health Organization (WHO) classification.
  For example:hematotoxicity,nausea,fatigue, abnormal liver function, alopecia, peripheral nerve damage, and constipation et al.
Overall response rate (ORR) | 2 years
  The disease control rate,This is the equivalent to Overall response rate, was (CR+ PR+SD).CR:complete respons; PR:partial response; SD:stable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Wang, master, Study Director — Study Director

REFERENCES:
- [Result] Raizer JJ, Rademaker A, Evens AM, Rice L, Schwartz M, Chandler JP, Getch CC, Tellez C, Grimm SA. Pemetrexed in the treatment of relapsed/refractory primary central nervous system lymphoma. Cancer. 2012 Aug 1;118(15):3743-8. doi: 10.1002/cncr.26709. Epub 2011 Dec 16. PMID 22179954
- [Result] Zhang JP, Lee EQ, Nayak L, Doherty L, Kesari S, Muzikansky A, Norden AD, Chen H, Wen PY, Drappatz J. Retrospective study of pemetrexed as salvage therapy for central nervous system lymphoma. J Neurooncol. 2013 Oct;115(1):71-7. doi: 10.1007/s11060-013-1196-1. Epub 2013 Jul 5. PMID 23828279
- [Result] Leshchenko VV, Kuo PY, Jiang Z, Thirukonda VK, Parekh S. Integrative genomic analysis of temozolomide resistance in diffuse large B-cell lymphoma. Clin Cancer Res. 2014 Jan 15;20(2):382-92. doi: 10.1158/1078-0432.CCR-13-0669. Epub 2013 Oct 31. PMID 24178621